CLINICAL TRIAL: NCT03107507
Title: Efficacy of Levetiracetam in Control of Neonatal Seizures
Brief Title: Efficacy of Levetiracetam in Control of Neonatal Seizures Guided by an EEG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Salah Shaheen, Pricipal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YSShaheen
Record Dates: First submitted 2017-02-22; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Neonatal Seizures
Keywords: EEG with Periodic Abnormalities; Levetiracetam; Phenobarbitone; neonatal seizures; Neurodevelopmental Abnormality
MeSH Terms: interventions — Levetiracetam; Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam (Active Comparator): Levetiracetam given in oral form via oro-gastric tube, first a bolus dose 40-50mg/kg then maintenance dose 10-30 mg/kg/day divided every 12 hours.
  Duration: until seizure free
  Interventions: Drug: Levetiracetam
- Phenobarbital (Active Comparator): Phenobarbital given in IV form, loading dose 20mg/kg that can be repeated after a 20 minute interval not to exceed 40mg/kg then maintenance dose 2-4 mg/kg/day divided every 12 hours.
  Duration: until seizure free
  Interventions: Drug: Phenobarbital

INTERVENTIONS:
Drug: Levetiracetam — Given in a bolus dose first 50mg/kg as levetiracetam reaches a therapeutic serum level rapidly in 1.3 hours. Titration will not be attempted in our study to reach drug level rapidly and consequent rapid effective control of seizures. Maintenance dose is then given at a dose of 10 - 40mg/kg/day divided every 12 hours.
  Arms: Levetiracetam
Drug: Phenobarbital — Phenobarbital is given intravenously in the form of a loading dose of 15mg/kg that can be repeated after a 20 minute interval not to exceed 30mg/kg then a maintenance dose 2-4 mg/kg/day divided every 12 hours.
  Arms: Phenobarbital

SUMMARY:
Over the last three decades, several tools have been developed to enhance the detection and treatment of neonatal seizures. Regarding treatment, phenobarbital maintains is still used as a first-line therapy worldwide. However, newer anti-epileptic drugs (AED) s such as, levetiracetam, bumetanide, and topiramate are increasingly being applied to the neonatal population, offering the potential for seizure treatment with a significantly better side-effect profile.

Levetiracetam is a very promising medication for the treatment of neonatal seizures. It has been in clinical use for almost a decade in adults and older children with good efficacy, an excellent safety profile and near ideal pharmacokinetic characteristics. It has been approved and used for treatment of seizures in infants starting one month of age since 2012.

The investigators are comparing the efficacy of levetiracetam to that of phenobarbital as a first-line drug in control of neonatal seizures. The investigators monitor the efficacy through assessment of frequency of seizures before and after drug administration, amplitude integrated EEG changes in background activity and seizure frequency in participants, duration taken for participants to be seizure free and short term neurodevelopmental outcome and EEG at 3 months of age

ELIGIBILITY:
Inclusion Criteria:

* All full term neonates experiencing seizures due to; post-hypoxic or post-ischemic encephalopathy, intracerebral hemorrhage, cerebral infection, inborn errors of metabolism or malformations of cortical development

Exclusion Criteria:

* Preterm neonates
* Full term neonates with seizures due to metabolic derangements (hypoglycemia, hypocalcemia or hypomagnesemia)
* Full term neonates with impaired renal functions.

Ages: 1 Hour to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-03-25 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of levetiracetam in control of neonatal seizures as a first line versus phenobarbital through assessment of seizure burden. | 72 hours
  Number of seizures before and after levetiracetam administration in comparison to phenobarbital.
Efficacy of levetiracetam in rapid control of neonatal seizures compared to phenobarbital. | 72 hours
  Number of hours taken to achieve seizure freedom after administration of levetiracetam versus phenobarbital.

SECONDARY OUTCOMES:
Dose escalation data about levetiracetam through studying the efficacy of further dose administration in non responders. | 72 hours
  Number of originally non responder participants who achieved seizure control with higher doses of levetiracetam.
Adequacy of levetiracetam as a single agent antiepileptic drug in control of neonatal seizures. | 30 days
  Number of participants who require addition of second line antiepileptic drug to control seizures after levetiracetam versus phenobarbital use.
Accuracy of amplitude integrated EEG monitoring in detecting neonatal seizures before and after antiepileptic drug use. | 48 hours
  Number of seizures detected by aEEG before and after antiepileptic drug use.
Effect of levetiracetam on aEEG background activity of participants. | 48 hours
  Number of participants with normalization of background activity after administration of levetiracetam versus phenobarbital.
The short term clinical outcome of patients with neonatal seizures after treatment with levetiracetam. | 3 months
  Neurodevelopmental assessment through detecting presence of following milestones:
  1. Head control
  2. Social smile
  3. Visual fixation and pursuit
  4. Turning towards sounds
The short term electroencephalographic outcome of patients with neonatal seizures after treatment with levetiracetam | 3 months
  Number of participants with presence of epileptogenic activity on follow up electroencephalogram.

OTHER OUTCOMES:
To gather safety information on levetiracetam use in neonates | 72 hours
  By collecting data of renal and liver function tests 48-72 hours after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Omneya G Afify, MD, Study Chair — Cairo University; Iman F Iskander, MD, Study Director — Cairo University; Aliaa A Ali, MD, Principal Investigator — Cairo University; Yara S Shaheen, MSc., Principal Investigator — Cairo University; Walaa Shaarany, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Children's Hospital (Abulreesh), Cairo Governorate, Egypt